CLINICAL TRIAL: NCT06246591
Title: Extracorporeal Shockwave Therapy vs Mesotherapy in the Treatment of Myofascial Pain Syndrome: a Case-control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MFR012024
Record Dates: First submitted 2024-01-17; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Myofascial Pain Syndrome; Trigger Point Pain, Myofascial
Keywords: Muscle contracture; ESWT; Mesotherapy; Myofascial syndrome; Trigger point
MeSH Terms: conditions — Myofascial Pain Syndromes; Contracture | interventions — Extracorporeal Shockwave Therapy; Mesotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal Shockwave Therapy (Group A) (Active Comparator): Patients of this group were invited to our department's outpatient clinics on a weekly basis, for a total of five sessions (5 weeks), lasting approximately 20 minutes each. Treatment energy and frequency were established following the recommendations and guidelines of the International Society for Medical Shockwave Treatment (ISMST).
  Interventions: Other: Extracorporeal Shockwave Therapy (Group A)
- Mesotherapy (Group B) (Active Comparator): Patients in this group underwent mesotherapy treatment at our outpatient clinics with Thiocolchicoside fl 4mg/2ml and Mepivacaine fl 10mg/1ml, once a week, for a total of five sessions (5 weeks), lasting about 15 minutes each.
  Interventions: Other: Mesotherapy (Group B)

INTERVENTIONS:
Other: Extracorporeal Shockwave Therapy (Group A) — Each patient was evaluated before treatment for trigger points; patients underwent focal ESWT (PulseWave 2 - Mectronic Medicale s.r.l.) with a specific program for muscle contractures and myofascial pain (80-100 mJ with 2250 pulses of 5-10 Hz).
  Arms: Extracorporeal Shockwave Therapy (Group A)
Other: Mesotherapy (Group B) — Each patient was evaluated before treatment for trigger points; after disinfection with Chlorhexidine 2% and sterile gauze, Thiocolchicoside fl 4mg/2ml, and a local anesthetic, Mepivacaine fl 10mg/1ml, diluted in 0.9% NaCl saline, for a final volume of 10 ml, were inoculated mesodermally; 6 to 12 microinjections with needle 26G 0.40x4mm, were performed.
  Arms: Mesotherapy (Group B)

SUMMARY:
Myofascial Pain Syndrome (MPS) is a disorder of the musculoskeletal system manifested by referred pain associated with functional limitation, muscle contractures, and possible neuralgic manifestations; this condition is characterized by the presence of "trigger points". The goal of this case-control study was to compare the effects and benefits of treatment with ESWT vs Mesotherapy in myofascial pain syndrome. The main question it aims to answer is: what is the best rehabilitation project-program between ESWT and mesotherapy for patients with myofascial syndrome? A case-control study was conducted at the U.O.C. of "Recovery and Functional Rehabilitation" A.O.U.P. "P. Giaccone" of Palermo from February 2022 to Dicember2023. Patients were randomized into 2 groups: in group "A", No. 5 sessions of focal ESWT were given weekly; in group "B", No. 5 sessions of Mesotherapy with administration of Thiocolchicoside fl 4mg/2ml and Mepivacaine fl 10mg/1ml were given weekly. Patients in group "A" and group "B" were evaluated at baseline (T0), after 5 sessions (T1) and one month after the end of treatment (T2). Researchers will compare patients treated with ESWT and patients performing mesotherapy to see if there are real differences in terms of pain reduction and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-65 years
* Diagnosis of myofascial syndrome
* NRS at T0 ≥ 4
* Written informed consent

Exclusion Criteria:

* Pregnant patients
* Patients with malignancies already diagnosed or in the process of diagnostic definition
* Coagulation disorders and/or therapy with anticoagulants
* Skin lesions and/or local infections
* Contraindications and/or allergies to the active ingredients of Mesotherapy.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Extent of pain: Numeric Rating Scale (NRS 0-10) | At the time of recruitment (T0). After 5 weeks from the start of treatment (T1). After 30 days from the end of treatment (T2).
  The NRS is a subjective scale that rates the extent of pain with a score between 0 and 10; a score of 10 corresponds to maximum pain.
Intensity o f pain: Pressure pain threshold (PPT 1-4) | At the time of recruitment (T0). After 5 weeks from the start of treatment (T1). After 30 days from the end of treatment (T2).
  PPT is defined as the minimum force applied to induce pain in the patient with myofascial pain syndrome. It has a score between 0 and 4; a score of 4 indicates maximum pain.

SECONDARY OUTCOMES:
Autonomy in activities of daily living: Barthel Index (BI 0-100) | At the time of recruitment (T0). After 5 weeks from the start of treatment (T1). After 30 days from the end of treatment (T2).
  BI is a scale that assesses the patient's autonomy in ADL. A score of 100 corresponds to a normal value.
Quality of life: Short Form Health Survey 36 (0-100) | At the time of recruitment (T0). After 5 weeks from the start of treatment (T1). After 30 days from the end of treatment (T2).
  SF-36 is a scale that assesses the quality of life in relation to the disease from which patients suffer. A score of 100 corresponds to an optimal value.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Letizia Mauro, Principal Investigator — Functional Recovery and Rehabilitation Unit of the A.O.U.P. Paolo Giaccone
Locations (1):
- Functional Recovery and Rehabilitation Unit of the A.O.U.P. Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Paoletta M, Moretti A, Liguori S, Toro G, Gimigliano F, Iolascon G. Efficacy and Effectiveness of Extracorporeal Shockwave Therapy in Patients with Myofascial Pain or Fibromyalgia: A Scoping Review. Medicina (Kaunas). 2022 Jul 28;58(8):1014. doi: 10.3390/medicina58081014. PMID 36013480
- [Background] Jun JH, Park GY, Chae CS, Suh DC. The Effect of Extracorporeal Shock Wave Therapy on Pain Intensity and Neck Disability for Patients With Myofascial Pain Syndrome in the Neck and Shoulder: A Meta-Analysis of Randomized Controlled Trials. Am J Phys Med Rehabil. 2021 Feb 1;100(2):120-129. doi: 10.1097/PHM.0000000000001493. PMID 32520797
- [Background] Nahomi Kuroda M, Thomaz de Aquino Nava G, Baldini Prudencio C, Affonso Paulo D, Peixouto I, Yoshi Moroshima M, de Almeida Lourenco M, Nogueira da Silva C, Mercia Pascon Barbosa A, Rodrigues Pedroni C. Effect of ischemic compressions versus extracorporeal shockwave therapy on myofascial trigger points: A protocol of a randomized controlled trial. PLoS One. 2023 Mar 30;18(3):e0283337. doi: 10.1371/journal.pone.0283337. eCollection 2023. PMID 36996078